CLINICAL TRIAL: NCT04314544
Title: A Phase III, Randomized, Double-Blind, Single-Dose, Placebo-Controlled Study to Demonstrate the Efficacy and Safety of Tildrakizumab in Subjects With Active Psoriatic Arthritis I (INSPIRE 1)
Brief Title: Efficacy and Safety of Tildrakizumab Compared to Placebo in Subjects With Active Psoriatic Arthritis I (INSPIRE 1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TILD-19-07
Record Dates: First submitted 2020-03-13; First posted 2020-03-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Active Psoriatic Arthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: TILD
- Arm B (Placebo Comparator)
  Interventions: Drug: matching placebo injections

INTERVENTIONS:
Drug: TILD — one 1 mL injection of study medication
  Arms: Arm A
Drug: matching placebo injections — one 1 mL injection of placebo
  Arms: Arm B

SUMMARY:
This is a multicenter Phase III, Randomized, Double-Blind, Single-Dose, Placebo-Controlled Study to Demonstrate the Efficacy and Safety of tildrakizumab in Subjects with Active Psoriatic Arthritis I (INSPIRE 1)

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent.
2. Subject is ≥ 18 years of age at time of Screening.
3. RF and anti-CCP Ab negative.
4. Subjects must have prior exposure to anti-TNF agent(s) use for the treatment of PsO or PsA.

Exclusion Criteria:

1. Subject has a planned surgical intervention between Baseline and the Week 24 evaluation for a pretreatment condition.
2. Subject has an active infection or history of infections as follows:

   * any active infection for which systemic anti-infectives were used within 28 days prior to first IMP dose, with the last dose having been received within 7 days of Screening,
   * a serious infection, defined as requiring hospitalization or IV anti-infectives within 8 weeks prior to the first IMP dose, with the last dose having been received within 7 days of Screening,
   * recurrent or chronic infections, e.g., chronic pyelonephritis, chronic osteomyelitis, bronchiectasis, or other active infection that, in the opinion of the Investigator, might cause this study to be detrimental to the subject.
3. Subject has a known history of infection with hepatitis B, hepatitis C, or human immunodeficiency virus.
4. Subject had myocardial infarction, unstable angina pectoris, or ischemic stroke within the past 6 months prior to the first IMP dose.
5. Subject has any active malignancy, including evidence of cutaneous basal or squamous cell carcinoma or melanoma.
6. Subject has a history of malignancy within 5 years from the time of Screening EXCEPT treated and considered cured cutaneous basal or squamous cell carcinoma, in situ cervical carcinoma, OR in situ breast ductal carcinoma.
7. Subjects with a history of alcohol or drug abuse in the previous 2 years.
8. Female subjects of childbearing potential who do not agree to abstain from heterosexual activity or practice a dual method of contraception, for example, a combination of the following: (1) oral contraceptive, depo progesterone, or intrauterine device; and (2) a barrier method (condom or diaphragm). Male subjects with female partners of childbearing potential who are not using birth control as described above must use a barrier method of contraception (e.g., condom) if not surgically sterile (i.e., vasectomy). Contraceptive methods must be practiced upon entering the study and through 17 weeks after the last dose of IMP. If a subject discontinues prematurely, the contraceptive method must be practiced for 17 weeks following final administration of IMP. A FSH test should be performed to confirm menopause for those women with no menses for less than 1 year.
9. Subject currently enrolled in another investigational device/procedure or drug study, or Baseline of this study is less than 30 days or 5 half-lives (whichever is longer) since ending another investigational device/procedure or drug study(s), or receiving other investigational agent(s).
10. Subject previously has been enrolled (randomized) in this study.
11. Subject has any kind of disorder that, in the opinion of the Investigator, may compromise the ability of the subject to give written informed consent and/or to comply with all required study procedures.
12. Donation or loss of 400 mL or more of blood within 8 weeks before dosing.
13. Subjects who have been placed in an institution on official or judicial orders.
14. Subjects who are related to or dependent on the Investigator, Sponsor, or study site such that a conflict of interest could arise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-12-22 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who achieve American College of Rheumatology [ACR20] | at week 24
  the proportion of subjects achieving a 20% reduction from Baseline in response criteria

SECONDARY OUTCOMES:
The proportion of subjects achieving American College of Rheumatology [ACR50] | at Week 24
  the proportion of subjects achieving a 50% reduction from Baseline in response criteria
The proportion of subjects achieving American College of Rheumatology [ACR70] | at Week 24
  the proportion of subjects achieving a 70% reduction from Baseline in response criteria
The proportion of subjects achieving Psoriasis Area and Severity Index 75 response among subjects with Body surface area ≥3% at baseline | at Weeks 24
The change from Baseline in the van der Heijde modified total Sharp score | at Week 24
The change from Baseline in the van der Heijde modified total Sharp score | at Week 16
Change from Baseline in American College of Rheumatology Response Criteria Components Score | at Week 24
  Tender Joint Count (68), Swollen Joint Count (66), Physician's Global Assessment of Arthritis (Visual Analog Scale, 0-100), Patient's Global Assessment of Arthritis (Visual Analog Scale, 0-100), Patient's Assessment of Arthritis Pain (Visual Analog Scale, 0-100), C-reactive protein levels, Erythrocyte sedimentation rate levels
change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index | at Week 24
change from Baseline in Leeds Enthesitis Index | at Week 24
The change from Baseline in Leeds Dactylitis Index | at Week 24
The proportion of subjects who achieve a disease activity score-C-reactive protein < 3.2 | at Week 24
The change from Baseline in van der Heijde modified Sharp sub-scores (erosion score and joint space narrowing score) | at Week 24
The proportion of subjects with the Change in van der Heijde modified total Sharp score <0 and < 0.5 | at Week 24.
The proportion of subjects with active Psoriasis and Body surface area ≥3% | at Week 24
  with: Psoriasis Area and Severity Index 90 and Psoriasis Area and Severity Index 100
The change from Baseline in subjects with active Psoriasis and Body surface area ≥ 3% ("those with involvement of nails" ) | at Week 24
  Physician Global Assessment-Psoriasis and nail psoriasis severity index
The proportion of subjects achieving American College of Rheumatology [ACR20, ACR50 and ACR70] | at week 52
  the proportion of subjects achieving a 20/50/70% reduction from Baseline in response criteria
The change from Baseline in American College of Rheumatology Response Criteria Components Score | at Week 52
  Tender Joint Count (68), Swollen Joint Count (66), Physician's Global Assessment of Arthritis (Visual Analog Scale, 0-100), Patient's Global Assessment of Arthritis (Visual Analog Scale, 0-100), Patient's Assessment of Arthritis Pain (Visual Analog Scale, 0-100), C-reactive protein levels, Erythrocyte sedimentation rate levels
The change from Baseline in Bath Ankylosing Spondylitis Disease Activity Index | at Week 52
The change from Baseline | at Week 52
  Leeds Enthesitis Index, Leeds Dactylitis Index, Health Assessment Questionnaire Disability Index Score
The proportion of subjects who achieve a Disease Activity Score(28 [joints]-C-reactive protein) < 3.2 | at Week 52
The change from Baseline in van der Heijde modified total Sharp score | at Week 52
The change from Baseline in van der Heijde modified Sharp sub-scores (erosion score and joint space narrowing score) | at Week 52
The proportion of subjects with the change in van der Heijde modified total Sharp score <0 and < 0.5 | at Week 52
In subjects with active Psoriasis and Body surface area ≥3%, the proportion of subjects | at Week 52
  Psoriasis Area and Severity Index 75, Psoriasis Area and Severity Index 90 and Psoriasis Area and Severity Index 100
In subjects with active Psoriasis and Body surface area ≥3% those with involvement of nails , the change from Baseline in nail psoriasis severity index | at Week 52
In subjects with active Psoriasis and Body surface area ≥3%, the change from Baseline in Physician Global Assessment-Psoriasis | at Week 52
Change from baseline in health assessment questionnaire - disability index (HAQ-DI) score | at Week 24
The change from Baseline in the Short-Form-36 Health Survey Version 2 (SF-36v2), Acute Components | Weeks 24 and 52
  Physical Functioning Domain, Role-Physical Domain, Role-Emotional Domain, Bodily Pain Domain, Mental Health Domain, General Health Domain, Vitality Domain, Social Functioning Domain, Physical Component Summary Score, Mental Component Summary Score
The change from Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue Scores | at Week 24

OTHER OUTCOMES:
The proportion of subjects achieving American College of Rheumatology [ACR20] | Weeks 24 and 52
  the proportion of subjects achieving a 20% reduction from Baseline in response criteria
The proportion of subjects achieving American College of Rheumatology [ACR50] | Weeks 24 and 52
  the proportion of subjects achieving a 50% reduction from Baseline in response criteria
The proportion of subjects achieving American College of Rheumatology [ACR70] | Weeks 24 and 52
  the proportion of subjects achieving a 70% reduction from Baseline in response criteria
The change from Baseline in American College of Rheumatology Response Criteria Components Score | Weeks 24 and 52
  Tender Joint Count (68), Swollen Joint Count (66), Physician's Global Assessment of Arthritis (Visual Analog Scale, 0-100), Patient's Global Assessment of Arthritis (Visual Analog Scale, 0-100), Patient's Assessment of Arthritis Pain (Visual Analog Scale, 0-100), C-reactive protein levels and Erythrocyte sedimentation rate levels
The change from Baseline | Weeks 24 and 52
  Leeds Enthesitis Index, Leeds Dactylitis Index, Bath Ankylosing Spondylitis Disease Activity Index and Health Assessment Questionnaire Disability Index score
The proportion of subjects who achieve a Disease activity score-C-reactive protein < 3.2 | Weeks 24 and 52
The proportion of subjects with active Psoriasis and Body surface area ≥ 3% | Weeks 24 and 52
  Psoriasis Area and Severity Index 75, Psoriasis Area and Severity Index 90 and Psoriasis Area and Severity Index 100
The change from Baseline in the levels of "Metabolic Biomarkers" | at Week 24
the change from baseline in Disease Activity Index for Psoriatic Arthritis (DAPSA) | at Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and Week 52
proportion of subjects who achieve a response based on Modified Psoriatic Arthritis Responder Criteria (PsARC) | at Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and Week 52.
change from baseline in Work Productivity and Activity Impairment Questionnaire Scores | at Week 12,16 24, 48 and 52
change from baseline in Psoriatic Arthritis Disease Activity Score (PASDAS) | at Week 8,16, 24 and 52.

CONTACTS AND LOCATIONS:
Locations (97):
- United States (45):
  - Sunpharma Site no 42, Dothan, Alabama
  - Sunpharma Site no 29, Gilbert, Arizona
  - Sunpharma Site no 30, Glendale, Arizona
  - Sunpharma Site no 31, Mesa, Arizona
  - Sunpharma Site no 35, Covina, California
  - Sunpharma Site no 48, Encino, California
  - Sunpharma site no. 17, Fountain Valley, California
  - Sunpharma site no. 15, Thousand Oaks, California
  - Sunpharma Site no. 141, Avon Park, Florida
  - Sunpharma site no. 21, Clearwater, Florida
  - Sunpharma site no. 02, Hialeah, Florida
  - Sunpharma Site no 55, Kissimmee, Florida
  - Sunpharma Site no. 75, Margate, Florida
  - Sunpharma site no. 05, New Port Richey, Florida
  - Sunpharma Site no. 76, Ocoee, Florida
  - SunPharma Site no 22, Tamarac, Florida
  - Sunpharma Site no 46, Gainesville, Georgia
  - Sunpharma Site no 41, Oak Brook, Illinois
  - Sunpharma Site no 54, Orland Park, Illinois
  - Sunpharma Site no 38, Schaumburg, Illinois
  - Sunpharma Site no 37, Skokie, Illinois
  - Sunpharma Site no. 122, Skokie, Illinois
  - Sunpharma site no. 20, Wichita, Kansas
  - Sunpharma site no. 07, Worcester, Massachusetts
  - Sunpharma site no. 14, Springfield, Missouri
  - Sunpharma Site no 53, Kalispell, Montana
  - Sunpharma Site no 27, Lincoln, Nebraska
  - Sunpharma Site no 44, Voorhees Township, New Jersey
  - Sunpharma Site no 52, Charlotte, North Carolina
  - Sunpharma Site no. 73, Leland, North Carolina
  - Sunpharma Site no 56, Wilmington, North Carolina
  - Sunpharma Site no 33, Minot, North Dakota
  - Sunpharma site no. 11, Middleburg Heights, Ohio
  - Sunpharma Site no. 124, Oklahoma City, Oklahoma
  - Sunpharma Site no 34, Greenville, South Carolina
  - Sunpharma Site no 50, Austin, Texas
  - Sunpharma site no. 13, Baytown, Texas
  - Sunpharma Site no 49, Colleyville, Texas
  - Sunpharma site no. 08, Houston, Texas
  - Sunpharma Site no 28, Lubbock, Texas
  - Sunpharma Site no. 74, Mesquite, Texas
  - Sunpharma site no. 16, San Antonio, Texas
  - Sunpharma Site no 26, Stafford, Texas
  - Sunpharma site no. 01, Tomball, Texas
  - Sunpharma Site no. 121, Salt Lake City, Utah
- Sunpharma site 98, Trois-Rivières, Quebec, Canada
- Czechia (4):
  - Sun pharma site 99, Brno
  - Sunpharma Site no. 100, Prague
  - Sunpharma Site no. 101, Prague
  - Sunpharma Site no. 96, Zlín
- Estonia (3):
  - Sunpharma Site no. 85, Tallinn
  - Sunpharma Site no. 87, Tartu
  - Sunpharma Site no. 86, Tartu
- Germany (2):
  - Sunpharma Site no. 91, Berlin
  - Sunpharma Site no. 103, Herne
- India (10):
  - Sunpharma Site no. 128, Mylapore, Chennai
  - Sunpharma Site no. 134, Surat, Gujarat
  - Sunpharma Site no. 127, Bangalore, Karnataka
  - Sunpharma Site no. 130, Belagavi, Karnataka
  - Sunpharma Site no. 132, Hubli, Karnataka
  - Sunpharma Site no. 143, Kochi, Kerala
  - Sunpharma Site no. 131, Pune, Maharashtra
  - Sunpharma Site no. 142, Pune, Maharashtra
  - Sunpharma Site no. 129, Lucknow, Uttar Pradesh
  - Sunpharma Site no. 144, Kolkata, West Bengal
- Italy (2):
  - Sunpharma Site no. 104, Milan
  - Sunpharma Site no. 138, Verona
- Poland (12):
  - Sunpharma Site no. 95, Warsaw, Mazowiecki
  - Sunpharma Site no. 110, Bialystok
  - Sunpharma Site no. 93, Bialystok
  - Sunpharma Site no. 139, Katowice
  - Sunpharma Site no. 94, Krakow
  - Sunpharma Site no. 107, Lublin
  - Sunpharma Site no. 136, Olsztyn
  - Sunpharma Site no. 106, Ponzan
  - Sunpharma Site no. 92, Poznan
  - Sunpharma Site no. 108, Torun
  - Sunpharma Site no. 111, Warsaw
  - Sunpharma Site no. 137, Wroclaw
- Slovakia (2):
  - Sunpharma Site no. 88, Martin
  - Sunpharma Site no. 112, Vahom
- South Korea (2):
  - Sunpharma Site no 71, Seoul
  - Sunpharma Site no 70, Seoul
- Spain (8):
  - Sunpharma Site no 58, A Coruña
  - SunPharma Site No 23, Córdoba
  - Sunpharma Site no. 78, Madrid
  - Sunpharma Site no. 116, Málaga
  - Sunpharma Site no. 125, Sabadell
  - Sunpharma Site no. 115, Santiago de Compostela
  - Sunpharma Site no. 117, Seville
  - Sunpharma Site no 59, Valencia
- Taiwan (6):
  - Sunpharma Site no 65, Taipei, Pai-Tou
  - Sunpharma Site no 63, Jianguo, Taichung
  - Sunpharma Site no. 79, Hsinchu
  - Sunpharma Site no 62, Kaohsiung City
  - Sunpharma Site no 60, Tainan
  - Sunpharma Site no 64, Taipei

IPD SHARING:
Plan to Share IPD: No